CLINICAL TRIAL: NCT06324825
Title: Fuzhegn Nizeng Formula for Chronic Atrophic Gastritis With Low-grade Intraepithelial Neoplasia, a Multicenter Randomized Controlled Trial
Brief Title: Fuzheng Nizeng Formula for Chronic Atrophic Gastritis With Low-grade Intraepithelial Neoplasia, a Multicenter Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022CR64
Record Dates: First submitted 2023-09-01; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Atrophic Gastritis With Low-grade Intraepithelial Neoplasia
Keywords: Atrophic Gastritis; Intraepithelial Neoplasia
MeSH Terms: conditions — Gastritis, Atrophic; Carcinoma in Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fuzhegn Nizeng Formula (Experimental)
  Interventions: Drug: Fuzhegn Nizeng Decoction
- Moluodan patient medicine (Active Comparator)
  Interventions: Drug: Moluodan granules

INTERVENTIONS:
Drug: Fuzhegn Nizeng Decoction — Subjects taking prepared Fuzhegn Nizeng granules twice daily for 6 month.
  Arms: Fuzhegn Nizeng Formula
Drug: Moluodan granules — Subjects taking prepared Moluodan granules 9g twice daily for 6 month.
  Arms: Moluodan patient medicine

SUMMARY:
Fuzheng Nizeng Formula (FZNZ) is derived from the classic formula Liujunzi Decoction. Former pilot study found that FZNZ promoted the recovery of gastric atrophy and relieve the relative symptoms. This study is to evaluate its efficacy for chronic atrophic gastritis with low-grade intraepithelial neoplasia, compared with positive control Molduodan granule.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Atrophic Gastritis With Low-grade Intraepithelial Neoplasia diagnosed by endoscopy and stomach biopsy.
* Helicobacter pylori negative.
* TCM syndrome is spleen-stomach deficiency with blood stasis and phelgm.

Exclusion Criteria:

* History of gastric surgery.
* Combined with malignant tumor.
* History of mental illness.
* Allergy to any components of the drug use in the study.
* Planning to pregnancy, or pregnant woman and lactating woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Recovery rate of Low-grade Intraepithelial Neoplasia | The 180 days after drug administration.
  Stomach biopsy will be taken after drug administration completion.

SECONDARY OUTCOMES:
7-point Global Overall Symptom Scale | 1st, 2nd, 3rd, 4th, 5th, 6th month
  Dyspepsia symptoms will be recorded and evaluated by 7-point Global Overall Symptom Scale
Adverse event rate | The 6 months during the drug administration
  Any adverse event will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided